CLINICAL TRIAL: NCT04530799
Title: Influenza-associated Pulmonary Aspergillosis (IAPA) in ICU Patients With Severe Influenza: Incidence and Host- and Pathogen Related Risk Factors
Brief Title: Prospective Observational Trial of IAPA
Acronym: IAPAFLU
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IAPAFLU
Record Dates: First submitted 2020-08-20; First posted 2020-08-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Influenza With Pneumonia; Pulmonary Aspergillosis
Keywords: Influenza; Intensive Care Unit; Influenza-associated pulmonary aspergillose; Invasive Pulmonary Aspergillosis; Virus Diseases; Respiratory tract infections; Fungal Lung Diseases
MeSH Terms: conditions — Pulmonary Aspergillosis; Influenza, Human; Invasive Pulmonary Aspergillosis; Virus Diseases; Respiratory Tract Infections; Lung Diseases, Fungal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IAPA+: Influenza patients who develop IAPA during ICU admission
  Interventions: Other: Identification of biomarkers for IAPA via patient sampling
- IAPA-: Influenza patients admitted to the ICU not developing IAPA
  Interventions: Other: Identification of biomarkers for IAPA via patient sampling

INTERVENTIONS:
Other: Identification of biomarkers for IAPA via patient sampling — Blood, BAL, microbiome

SUMMARY:
A prospective multi-center observational study to assess the incidence of influenza-associated pulmonary aspergillosis (IAPA) in ICU patients and to identify host- and pathogen related risk factors for IAPA in EORTC negative ICU patients with severe influenza.

DETAILED DESCRIPTION:
Invasive pulmonary aspergillosis was shown to be a complication of severe influenza infections in immunocompromised patients as well as in immunocompetent patients and is associated with a high mortality. Antifungal prophylaxis might prevent influenza-associated pulmonary aspergillosis (IAPA) and thus might improve the outcome in patients with severe influenza. However, clinical related risk factors should be identified to assess whether a patient will benefit from antifungal prophylaxis. This prospective multi-center observational study will assess the incidence of influenza-associated pulmonary aspergillosis (IAPA) in ICU patients in 12 ICUs in The Netherlands, Belgium and France over 4 influenza seasons. The secondary objective of this study is to identify host- and pathogen related risk factors for IAPA in EORTC negative ICU patients with severe influenza. Patients aged 18 or older admitted to the intensive care unit (ICU) during the inclusion period due severe influenza without classic risk factors defined by the EORTC will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PCR-positive respiratory virus panel (RVP) result for influenza within 96 hours before or 48 hours after ICU admission.
* Patients who require ICU admission for more than 24 hours for severe influenza.
* Patients who have respiratory distress (respiratory rate >= 25x/minute and paO2/fiO2 < 300 with or without bilateral infiltrates) as the main reason for ICU admission.
* Patients who do not have an EORTC host factor.
* Patients who are at least 18 years of age.

Exclusion Criteria:

* Patients with age < 18 years as extensive sampling is required
* Expected survival on ICU admission ≤ 48h
* Patients that are being treated actively with antifungal agents for invasive aspergillosis.
* Patients or their legal representatives who did not sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target patient population is the EORTC-negative population of critically ill influenza patients at ICU. Patient identification will rely on daily review of ICU patients with respiratory virus panels ordered in the previous 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of IAPA-infection at ICU discharge | from date of admission in ICU assessed up to ICU discharge, approximately 21 days
  The diagnosis of IAPA will be made by the treating physician, according to a strict case definition.

SECONDARY OUTCOMES:
Time to IAPA diagnosis | from date of admission in ICU assessed up to ICU discharge, approximately 21 days
  The diagnosis of IAPA will be made by the treating physician, according to a strict case definition.
Length of ICU stay | from date of admission in ICU assessed up to ICU discharge, approximately 21 days
Length of hospital stay | from date of admission in hospital assessed up to hospital discharge, approximately 30 days
ICU mortality | up to ICU discharge, approximately 21 days
Hospital mortality | from date of admission in hospital assessed up to hospital discharge, approximately 30 days
30-day mortality | 30 days
90-day mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Joost Wauters, MD, PhD, Principal Investigator — UZ Leuven
Locations (12):
- Belgium (3):
  - AZ St-Jan, Bruges
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- France (6):
  - Amiens-Picardie University Hospital, Amiens
  - Centre Hospitalier REgional Universitaire de Lille, Lille
  - Henri Mondor Hopital, Paris
  - Hopital Bichat, Paris
  - Hopital Lariboisiere, Paris
  - Hopital Pontchaillou, Centre Hospitalier Universitaire de Rennes, Rennes
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - AmsterdamUMC, locatie VUmc, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided